CLINICAL TRIAL: NCT03133364
Title: Developing and Testing Delicious and Nutritious for the Old People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Arne Astrup, Head of institute (Nutrition Exercise and Sports), University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-17002835
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Quality of Life; Nutritional Deficiency; Physical Performance
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: 2-armed randomized controlled study which in total runs 12 weeks.
  It has been calculated that 106 participants should be completed. With the risk of loss, 150 elderly are screened and invited to join the study, whereas 120 elderly should be included.
  Fifty participants are randomized to receive a control menu for 12 weeks and fifty participants are randomized to receive an intervention menu for 12 weeks.
  To enhance subject compliance and avoid treatment group contamination the randomization will be done in "blocks" where each of the 8 departments of the nursing home is randomized to either the Control or Intervention group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants are randomized to the control group (C) and intervention group (I) using the programme "Research randomizer". The main supervisor will manage the randomization.
  Participants are blinded to whether they receive the control or intervention menu. Each menu will daily consist of a main meal and a between-meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory optimized meals (Active Comparator): Intervention group is receiving:
  Popular dishes selected from hospital and meal service menus optimized by sensory experts. Optimization is done with respect to taste, texture and appereance and on nutritional composition of the meals with focus on protein content.
  Interventions: Other: Sensory optimized meals
- Control (Placebo Comparator): Control group is receiving:
  Popular dishes selected from hospital and meal service menus, NOT optimized by sensory experts.
  Interventions: Other: Sensory optimized meals

INTERVENTIONS:
Other: Sensory optimized meals — 19 main meals and 12 between-meals are optimized and composed to a menu for 12 weeks.

SUMMARY:
Meals-on wheels may play a major role in contributing to better nourishment and quality of life in older people, thus delaying costly hospitalisation. Still, dwelling, old adults who receive meals-on-wheels are a population at risk of undernutrition leading to a decreased quality of life.

Hypothesis Offering nutritious ELDORADO meals as meals-on-wheels to nursing home residents in 3 months is an effective way to increase quality of life.

Aim To improve quality of life and functional abilities in nursing home residents by offering nutritious ELDORADO meals.

DETAILED DESCRIPTION:
Intervention The intervention group (n=50) will receive an optimized menu (in both sensory and nutritious aspects) for 12 weeks. In cooperation with the Copenhagen house of food and sensory staff, 19 main meals and 12 between-meals have been optimized based on nursing home residents' evaluations of sensory aspects. On a daily basis the menu will consist of 1 optimized main meal and 1 optimized between-meal, served for dinner. There will be no selective choice for the elderly. If a participant does not want the daily meal, he will receive another meal from the ordinary menu from the kitchen.

Control In comparison, the control group (n=50) will receive the same menu as the intervention group, however, the meals are not optimized on sensory and nutritious aspects. On a daily basis this menu also includes 1 main meal and 1 between-meal in 12 weeks. If a participant does not want the daily meal, he will receive another meal from the ordinary menu from the kitchen.

ELIGIBILITY:
Inclusion Criteria:

* Living at Skovhuset, nursing home in Hillerød municipality, Denmark.
* Collecting the "energy-dense diet" "ældrekost" with 40 % fat, with a main meal and a dessert/starter.
* Able to understand and follow instructions for the procedures of the study.
* Above 65 years.

Exclusion Criteria:

* Have chewing or swallowing difficulties.
* Have acute disease or acute change in chronic disease.
* Living after special nutritional standards e.g. vegetarian, have any food allergies, or if a participant is excluding common foods from their diet because of other reasons.
* Not able or willing to give informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (EQ-5D-3L) | 12 weeks
  (EQ-5D-3L) is a standardized instrument for use as a measure of health outcome. The EQ-5D-3L descriptive system comprises the following 5 dimensions (5D): mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels (3L): no problems (1 point), some problems (2 points), extreme problems (3 points).
  This gives a total of 245 different health states, adding unconscious and dead.

SECONDARY OUTCOMES:
MMSE (mini mental status) | 12 weeks
  MMSE-test (mental function) MMSE is the most frequently used cognitive screening test, and has been developed with the aim of measuring cognitive abilities in the elderly and possibly changes in cognitive functioning over time.
Hand grip strenght | 12 weeks
  Hand Grip Strenght (HGS) is valid as a measure of mobility in both healthy people and patients and is associated with both physical (strenght of function) and mental (quality of life) aspects of the participant.
  HGS will be measured (in kg) with a Jamar 5030J1 Hydraulic Hand Dynanometer. It displays grip force up to 90 kg.
Chair stand | 12 weeks
  By means of the modified 30 seconds chair-stand. Participants are asked to fold their arms across their chest and to stand up and sit down on a chair, as many times as possible during 30 seconds. The seat should be a height of at least 43 cm. In the modified version the arm rests are used for assistance or safety.
Diet registration | 4 days
  In this study four days of diet registration will be done both in the intervention period and the control period on each participant to compare the energy and protein intake at the ordinary diet and at the project diet (intervention or control).
Satisfaction with food related life (SWFL) | 12 weeks
  SWFL consist of five items that can be measured independently, or grouped into a single dimension. The participants evaluate their degree of agreement, with five statements of answer possibilities (from disagree completely to agree completely), and a higher level means a better SWFL score.
Weight | 12 weeks
  The body weight of the participant is measured in the morning in the participants' home on a bathroom scale.
Height | 12 weeks
  Height will be measured with a folding ruler.
EVS | 12 weeks
  The Eating Validation Scheme (EVS) is a Danish nutritional assessment chart, used to assess nutritional intake and risk factors.
Liking | One month in the middle of the intervention
  During an evening meal participants will evaluate sensory parameters of the side course and the main meal (appearance, taste and texture) with the counseling of a research assistant.
  A 5-point hedonic scale ranging from 1 (dislike very much) to 5 (like very much) with the medium response either like or dislike was chosen.
Compliance | 12 weeks
  A compliance sheet (compliance-week-schedule) of each week will be done to register how many times of the week the participant has eaten the project meals and how many times they have eaten something else from the ordinal menu (due to dislike of the ordinal menu or other reasons).
Observations of meals | One month in the middle of the intervention
  In order to identify differences in the way the meal is handled and served an observational visit is done on the eight departments of the nursing home. The scheme includes six items:
  * Preparation of the dinner,
  * Tableware and serving,
  * Presentation of the dinner,
  * The food and side dishes,
  * The ambiance during dinner,
  * The role of the staff during dinner. Differences or coincidences from the observations will be found and used as background information to describe the meal situation.

CONTACTS AND LOCATIONS:
Overall Officials: Signe Loftager Okkels, Msc, Principal Investigator — The Nutrition Research Unit, Gentofte University hospital.
Locations (1):
- Skovhuset, nursing home, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
If other researchers are interested in the data, I am planning to share them after publication of the results.

REFERENCES:
- [Derived] Okkels SL, Dybdal DR, Pedersen RJ, Klausen TW, Olsen A, Beck AM, Bugel S. A culinary twist of a two-course meals-on-wheels menu in a cluster-randomized controlled trial influencing health-related quality of life in nursing home residents. Clin Nutr ESPEN. 2021 Jun;43:137-147. doi: 10.1016/j.clnesp.2021.02.002. Epub 2021 Mar 2. PMID 34024505